CLINICAL TRIAL: NCT00000584
Title: Transfusion-Transmitted Cytomegalovirus Prevention in Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 304; R01HL029883-04 (Other Grant/Funding Number: US NIH Grant Number)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2005-12

CONDITIONS: Blood Transfusion; Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Immunoglobulins

INTERVENTIONS:
Drug: immunoglobulins

SUMMARY:
To evaluate the capacity of intravenously administered cytomegalovirus (CMV)-immune globin (CMVIG) to immunize high risk premature infants against CMV infections.

DETAILED DESCRIPTION:
BACKGROUND:

Premature infants who require multiple blood transfusions have a 15-30 percent incidence of cytomegalovirus infections. Many of these infections result in severe disease, with a mortality of about 20 percent. In theory, the infection could be avoided by using blood and blood products exclusively from CMV antibody negative donors. The use of such blood is impractical because it would require the rejection of approximately 40 percent of all blood donors. Studies had suggested that passively acquired antibody could reduce the incidence of disease in exposed neonates. This provided the rationale for the use of passive immunization with hyperimmune globin in premature infants likely to require multiple transfusions. Lots of high titer CMV immune globulin suitable for intravenous administration were prepared using a technique of screening outdated blood bank plasma for units with high levels of antibody to CMV.

DESIGN NARRATIVE:

Randomized, double-blind. Subjects received either prophylactic CMVIG-intravenously or a placebo. Infants were followed for up to 12 weeks after discharge. Total sample size was expected to be 650.

The study completion date listed in this record was inferred from last publication listed in the Citations section of this study record.

ELIGIBILITY:
Neonates at high risk for transfusion-transmitted CMV infection. The neonates were either premature, of low birth weight, or had respiratory distress requiring the presence of an umbilical catheter.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1983-07; Study Completion 1988-06 (Actual)

REFERENCES:
- [Background] Snydman DR. Prevention of cytomegalovirus-associated diseases with immunoglobulin. Transplant Proc. 1991 Jun;23(3 Suppl 3):131-5, discussion 135. No abstract available. PMID 1648817
- [Background] Snydman DR, Werner BG, Meissner HC, Cheeseman SH, Schwab J, Bednarek F, Kennedy JL Jr, Herschel M, Magno A, Levin MJ, et al. Use of cytomegalovirus immunoglobulin in multiply transfused premature neonates. Pediatr Infect Dis J. 1995 Jan;14(1):34-40. doi: 10.1097/00006454-199501000-00007. PMID 7715987